CLINICAL TRIAL: NCT06047041
Title: Evidence-Informed Mental Health Prevention, Assessment, Collaboration, and Treatment in Middle Schools
Brief Title: Implementation Supports for Improving Identification and Delivery of School-based Mental Health Supports for Middle Schools Students
Acronym: E-IMPACTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: University of South Carolina (Other); University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Michael Lyons, PhD, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5320
Record Dates: First submitted 2023-09-01; First posted 2023-09-21 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-03

CONDITIONS: Mental Health Issue
Keywords: Schools; Adolescent Health

STUDY DESIGN:
Intervention Model Description: School-level randomization to treatment arm.
Who Masked: Outcomes Assessor
Masking Description: Assessors of schoolwide implementation outcomes (i.e., the School-Wide Evaluation Tool [SET] and the Individual Student Systems Evaluation Tool [ISSET]) will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EIS Only (Active Comparator): EIS Only (active comparator) condition schools involve technical assistance to support the implementation EIS.
  Interventions: Behavioral: EIS Only
- EIS + ECHO (Experimental): EIS + ECHO (experimental) condition involves all of the activities included in the "EIS Only" condition and will include enhanced implementation supports. Enhanced implementation supports involve 1) monthly collaborative learning ECHO sessions for school student support team staff to support implementation of EIS and evidence-based mental and behavioral health practices and 2) individual school teams will also receive follow-up supports to promote the implementation strategies presented during ECHO sessions.
  Interventions: Behavioral: EIS + ECHO

INTERVENTIONS:
Behavioral: EIS Only — The EIS Only Condition includes middle schools who have elected to implement the EIS. The EIS:
  * Is an online tool to that enables schools to identify students in need of additional mental or behavioral health support and provides recommendations for evidence-based practices.
  * Asks teachers and students to report on 7 areas of student social-emotional functioning
  * Facilitates schools' understanding of social-emotional student needs and recommended evidence-based practices at a variety of levels (e.g., school-, grade-, and individual-level).
  EIS Only Condition supports include:
  * Technical assistance professional development sessions to support the implementation of EIS and schoolwide practices related to identifying and supporting student mental health needs.
  * Individualized technical assistance for schools to support EIS implementation.
  Arms: EIS Only
Behavioral: EIS + ECHO — EIS + ECHO supports include supports from the EIS Only condition plus:
  * Monthly ECHO sessions for student support teams (SSTs; e.g., interdisciplinary groups of staff tasked to support student mental health). The ECHO experience involves:
    * Didactic training to support EIS implementation and effective identification and support of student mental and behavioral health needs.
    * Case-based learning and collaborative problem-solving related to EIS implementation and effective identification and support of student mental and behavioral health needs.
    * Collaboration with colleagues in schools that are also implementing the EIS.
    * Opportunities to consult with university faculty and content experts in school mental health.
  * Individualized SST coaching supports to facilitate the implementation of mental and behavioral health practices and strategies discussed during ECHO sessions.
  Arms: EIS + ECHO

SUMMARY:
This study will assess how different types of training and support influence the way that school staff understand, and respond to, the mental and behavioral health needs of middle school students. Researchers will work with middle schools using a developed screening system (called the Early Identification System; EIS) and compare how staff and student outcomes change when schools receive two different types of training and support: 1) standard onboarding/training versus 2) participating in professional learning communities and coaching.

DETAILED DESCRIPTION:
The "Evidence-Informed Mental health Prevention, Assessment, Collaboration, & Treatment in Middle Schools" (E-IMPACTS) project will evaluate how different implementation supports promote the ability of school staff to identify, and support, the mental and behavioral health needs of middle school students.

The project will involve researchers from the University of Virginia, University of Missouri, and University of South Carolina and middle schools (i.e., grades 6-8) that have elected to use a brief, universal tool, called the Early Identification System (EIS). The EIS assesses mental and behavioral health of students and connects these data to intervention recommendations. The EIS is a fully developed and validated tool that was developed to help school staff to identify, and address, the mental or behavioral health needs in their school building. The EIS system was developed as a low/no cost system to 1) be administered fully online and 2) present school staff with actionable next steps for supporting youth mental health needs.

Using a school-level randomized controlled trial (RCT) design, this project will test if/how two different types of implementation support changes 1) the way school staff use EIS recommended practices and 2) student outcomes. Half of schools in the RCT will receive standard implementation supports for using EIS. This treatment condition, called "EIS only", involves the existing technical assistance and on-boarding provided to any school already choosing to use EIS. Schools in the other treatment condition, called EIS+ECHO, will receive additional professional development and implementation support. This will involve participating in 1) online professional learning communities following the "Extension for Community Healthcare Outcomes" (ECHO) model and 2) follow-up coaching. The E-IMPACTS ECHO model (a) connects student support teams (e.g., interdisciplinary groups of school staff) across schools with each other and with content experts (e.g., university faculty specializing in school mental health) to collaboratively problem solve challenges they may be experiencing related to supporting student mental and behavioral health needs, and (b) provides schools with follow-up supports to facilitate the implementation of strategies discussed in ECHO sessions.

The purpose of the RCT is to determine the "value-added" of the EIS + ECHO, compared to the EIS alone (EIS Only) in Virginia, Missouri, and South Carolina middle schools located in rural areas or small suburbs/cities (i.e., an active comparison condition). Researchers hypothesize that, relative to EIS Only, the EIS + ECHO condition will be associated with greater improvements in: (a) student emotional/behavioral and academic outcomes, (b) staff knowledge, self-efficacy, and practice outcomes, and (c) school-level implementation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Public middle schools (must include grades 6-8) planning to implement the EIS
* Located in rural areas, towns, & suburbs / cities (NCES locales)
* All children attending the schools and staff employed by the schools are eligible for inclusion

Exclusion Criteria:

* Previous use of EIS (i.e., use of all screening data and intervention hub)
* <70% response rate on pre-intervention implementation of EIS

Ages: 10 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 21350 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in youth mental health measured by the Early identification System | 2 time points (over 9 months)
  De-identified, student-level behavioral data collected via the Early Identification System. The measure is a psychometrically validated mental and behavioral health screening system measuring domains including attention problems, internalizing problems, and externalizing problems.
Change in staff knowledge of evidence-based school mental health practices as measured by the Perceptions of Response To Intervention Skills Survey | 2 time points (over 9 months)
  Staff perceptions of the skills they possess related to evidence-based screening, monitoring, and intervention will be measured using a modified version of the Perceptions of Response To Intervention Skills Survey - Revised (PRSS; α > .90 for all factors). Response options range from not skilled (1) to very highly scaled (5).
Change in staff behaviors of evidence-based school mental health practices as measured by the Perceptions of Practices Survey | 2 time points (over 9 months)
  Perceptions of Practices Survey (PPS; Castillo et al., 2016) measures the extent to which schools implement evidence-based screening, intervention, and progress monitoring practices to support student mental health (α = .96 for the behavior factor; Marshall, 2016). Staff will indicate on a 5-point scale how frequently the practice occurred in their school.
Change in staff burnout as measured by the Maslach Burnout Inventory | 2 time points (over 9 months)
  Maslach Burnout Inventory (MBI; Maslach & Jackson, 1981). Measures staff experiences of emotional exasperation and fatigue. Staff will complete the emotional exhaustion factor from the MBI - Educators Survey (MBI-ES, α > .80; Wheeler et a., 2011). Response options range from never (0) to daily (6).
Change in schoolwide school mental health implementation outcomes as measured by the School-wide Evaluation Tool | 2 time points (over 9 months)
  The School-Wide Evaluation Tool (SET; Sugai et al., 2001) measure the implementation of evidence-based programs within a tiered system. The SET measures school-wide activities related to the implementation of school mental health systems, targeted interventions, and individualized interventions. A trained assessor will track implementation of evidence-based programs in both conditions.
Change in schoolwide school mental health implementation outcomes as measured by the Individual School-wide Evaluation Tool | 2 time points (over 9 months)
  The Individual Student Systems Evaluation Tool (ISSET; Debnam, Pas, & Bradshaw, 2012) measures the implementation of evidence-based programs within a tiered system. The ISSET measures foundations, targeted interventions, and individualized interventions. A trained assessor will track implementation in both conditions.

SECONDARY OUTCOMES:
Number of students with disciplinary referrals | 2 time points (over 12 months)
  De-identified data on school on student discipline referrals will be measured across treatment conditions.
Student grades | 2 time points (over 12 months)
  De-identified data on school on student academic achievement will be measured across treatment conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Lyons, Ph.D., Principal Investigator — University of Virginia
Locations (3):
- United States (3):
  - University of Missouri, Columbia, Missouri
  - University of South Carolina, Columbia, South Carolina
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No